CLINICAL TRIAL: NCT04000516
Title: The Effects of Early and Late Time-Restricted Feeding on Body Composition: an Effectiveness Trial in Sedentary Adults With Overweight and Obesity
Brief Title: The Effects of Early and Late Time-Restricted Feeding on Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Emily Dhurandhar, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2017-99
Record Dates: First submitted 2019-06-19; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Time Restricted Feeding
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group was asked to continue their usual eating schedule and pattern.
- Evening Fasters (EF) (Experimental): Evening fasters were asked to not consume food after 3 pm until the next morning.
  Interventions: Behavioral: Time restricted feeding
- Morning Fasters (MF) (Experimental): Morning fasters were asked to not consume food from the time they woke until 11 am.
  Interventions: Behavioral: Time restricted feeding

INTERVENTIONS:
Behavioral: Time restricted feeding — Restricting the eating window to about 8 hours a day, during waking hours.
  Arms: Evening Fasters (EF); Morning Fasters (MF)

SUMMARY:
A randomized controlled trial to determine the effectiveness of either morning or evening time-restricted feeding on body composition in sedentary, breakfast eating overweight and obese adults. Three parallel groups were assigned to either morning fasting (MF), evening fasting (EF), or a control group and asked to do the intervention for 6 weeks. Changes in body composition (change in weight, percent body fat percent, and percent lean body mass) are the primary outcome, and hunger and satiety ratings and physical activity are secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults that are currently habitual breakfast eaters, of overweight or obese BMI (BMI 25-35)

Exclusion Criteria:

* Participation in any weight-reduction program, weight-loss diet, or other special diet within the previous 3 months.
* Currently sedentary.
* Any highly restrictive dietary patterns.
* Currently consumes breakfast at least 5 times per week.
* Weight loss or gain of >5% of body weight in the past 6 months for any reason except post-partum weight loss.
* Currently taking medication that suppresses or stimulates appetite.
* Currently taking medication that requires eating with food in the morning, including NSAIDs.
* History of prior surgical procedure for weight control or liposuction.
* Current smoker or quit smoking less than 6 months prior.
* Individuals who do resistance training two or more days per week
* Any major disease, including:
* Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).
* Active or chronic infections, including self-reported HIV positivity and active tuberculosis.
* Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease (e.g., coronary artery bypass, percutaneous transluminal coronary angioplasty) in the past 6 months; New York Heart Association Functional Class >2 with respect to congestive heart failure; stroke or transient ischemic attack in the past 6 months. Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
* Active renal disease.
* Lung disease: chronic obstructive airway disease requiring use of oxygen.
* Diagnosed diabetes (type 1 or 2) .
* Uncompensated or uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in opinion of the investigators, would impede conduct of the trial or completion of procedures.
* Conditions or behaviors likely to effect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent clinic staff; another household member is a participant or staff member in the trial; unwilling to accept treatment assignment by randomization; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away from participating clinics before trial completed; unable to walk 0.25 mile in 10 minutes.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months.
* A recent or ongoing problem with drug abuse or addiction.
* Excessive alcohol intake, either acute or chronic, defined as any one of the following: 1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24-hr period in the past 12 months; or 3) other evidence available to clinic staff.
* Working the "night shift" or any work schedule that would interfere with normal eating patterns.
* Not willing to be randomized to any of the three experimental conditions.
* Pregnancy and childbearing: currently pregnant or less than 3 months post partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during study; unwilling to report possible or confirmed pregnancies promptly during the course of the trial; unwilling to take Qualtrics Screening Survey adequate contraceptive measures if potentially fertile.
* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Change in body fat percent | 6 weeks
  body fat percent at final visit- body fat percent at initial visit
Change in percent lean mass | 6 weeks
  lean mass percent at final visit - lean mass percent at initial visit
Change in body weight | 6 weeks
  body weight at final visit - body weight at initial visit

SECONDARY OUTCOMES:
Change in 24-hour physical activity energy expenditure (PAEE) | change after 3 weeks of intervention
  PAEE at week 3 of intervention - PAEE at baseline
Hunger measured by Visual Analog Scale (How Hungry do you feel now?) before breaking fast Day 2 | Day 2
  Hunger on day 2 of fasting pattern just before breaking fast, compared to hunger at that time in control group
Hunger measured by Visual Analog Scale (How Hungry do you feel now?) before breaking fast Day 42 | Day 42
  Hunger on Day 42 of fasting pattern just before breaking fast, compared to hunger at that time in control group

OTHER OUTCOMES:
Compliance with fasting | 6 weeks of intervention, daily from start to finish
  Percent of days during entire 6-week trial when fasting pattern was adhered to as recommended, recorded daily through the entire study.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Dhurandhar, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology and Sport Managment, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the study are accepted for publication, de-identified data will be uploaded to the ICSPR database. The protocol will be shared as supplementary material through the journal where the study if published, if allowed.
Supporting Information: Study Protocol
Time Frame: Within 6 months of publication.